CLINICAL TRIAL: NCT06900517
Title: The Efficacy of Salvia Officinalis Gel in the Treatment of Periodontitis by Monitoring Gingival Crevicular Fluid Volume and Interleukin 17 Concentration
Brief Title: The Efficacy of Salvia Officinalis Gel in the Treatment of Periodontitis CLINICAL TRIAL
Acronym: clinical
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Sarah Alrihaymee, Head of periodontic department, University of Baghdad
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1/3/2025
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: From each participant, two sites of periodontal pockets ( ≥ 5 mm ) were selected and randomly allocated to either the test site (treated with scaling and RSD with S. officinalis gel) or the control site (treated with scaling and RSD alone).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Other): will be treated with scaling and root planing alone
  Interventions: Dietary Supplement: Salvia officinalis Gel
- Test (Experimental): Will be treated by scaling and root plaing with the addition of Salvia officinalis Gel locally
  Interventions: Dietary Supplement: Salvia officinalis Gel

INTERVENTIONS:
Dietary Supplement: Salvia officinalis Gel — From each participant, two sites of periodontal pockets ( ≥ 5 mm ) were selected and randomly allocated to either the test site (treated with scaling and RSD with S. officinalis gel) or the control site (treated with scaling and RSD alone).
  Other Names: Scaling and root planing

SUMMARY:
From each participant, two sites of periodontal pockets ( ≥ 5 mm ) were selected and randomly allocated to either the test site (treated with scaling and RSD with S. officinalis gel) or the control site (treated with scaling and RSD alone).

DETAILED DESCRIPTION:
Background: Phytotherapy relies on the use of extracts derived from plants in pharmaceutical form. Herbal products have been effective in reducing periodontal diseases, as stated by many studies. Gingival crevicular fluid volume and concentrations of certain cytokines are precise and objective parameters in evaluating periodontitis treatment.

Aim of the study: Assessment of local application of Salvia officinalis (S. officinalis) gel as an adjunctive to scaling and root surface debridement (RSD) in the management of periodontitis.

Methods: A randomized clinical trial of split-mouth design for twenty-three subjects with periodontitis was assessed in this study. From each participant, two sites of periodontal pockets ( ≥ 5 mm ) were selected and randomly allocated to either the test site (treated with scaling and RSD with S. officinalis gel) or the control site (treated with scaling and RSD alone). A highly sensitive enzyme-linked immunosorbent assay (ELISA) was used to determine the concentration of interleukin 17 (IL-17) in gingival crevicular fluid (GCF).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis had at least 20 natural teeth, with probing pocket depth (PPD) ≥ 5 mm and attachment loss ≥ 4 mm

Exclusion Criteria:

* Exclusion criteria were pregnancy, lactation, smoking, and any systemic disease that might affect periodontal disease progression or require antibiotic usage. Likewise, patients who had received anti-inflammatory medications or antibiotics in the preceding three months were excluded.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
GCF volume | 1 month
  assessment the volume of GCF

SECONDARY OUTCOMES:
IL-17 | one month
  Assessment of IL-17